CLINICAL TRIAL: NCT04865913
Title: Venous Thrombosis Virtual Surveillance in COVID-19
Acronym: VVIRTUOSO
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 20200677-01T
Record Dates: First submitted 2021-04-27; First posted 2021-04-29 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Covid19; Venous Thromboembolism; Deep Vein Thrombosis; Pulmonary Embolism
MeSH Terms: conditions — COVID-19; Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational — A brief 15 min phone call 1 week, 30 and 90 days post discharge.

SUMMARY:
The overall goal of the VVIRTUOSO study is to determine the incidence of VTE including symptomatic DVT and PE after hospital discharge in patients with COVID-19 by implementing a pragmatic patient-centred prospective virtual VTE monitoring program in Canada and the United States.

DETAILED DESCRIPTION:
Emerging evidence suggests that COVID-19 induces a highly prothrombotic state particularly among hospitalized patients based on abnormal coagulation parameters and high rates of venous thromboembolism (VTE). Reported rates of VTE among hospitalized ward (3%) and critically ill (17% to 69%) patients with COVID-19 suggest that the risk of VTE is substantially higher than patients with other acute medical illnesses. VTE, which includes deep vein thrombosis (DVT) and pulmonary embolism (PE), is one of the most common preventable causes of hospital-associated morbidity and mortality, and most events occur after hospital discharge. The incidence of VTE after hospitalization for COVID-19 is not currently known. However, the combination of COVID-induced hypercoagulability, ongoing recovery, reduced mobility, advanced age, and comorbidities likely confers a high risk of VTE in this setting. The overall goal of the VVIRTUOSO study is to determine the incidence of VTE including symptomatic DVT and PE after hospital discharge in patients with COVID-19 by implementing a pragmatic patient-centred prospective virtual VTE monitoring program at 12 sites in Canada and the United States. Additional objectives are to explore risk factors for VTE post-discharge, characterize the use of pharmacological measures for VTE prevention, assess patient awareness of VTE and provide VTE education.

ELIGIBILITY:
Inclusion Criteria:

i) adults 18 years of age or older (or their delegate) ii) admitted to hospital with COVID-19 (laboratory confirmed) or diagnosed with COVID-19 (laboratory confirmed) during hospitalization iii) discharged from acute care hospital within prior 7 days.

Exclusion Criteria:

i) unconfirmed diagnosis of COVID-19, ii) no access to a telephone, computer or tablet for virtual assessment, iii) treated with therapeutic doses of anticoagulation after hospital discharge (e.g. atrial fibrillation, mechanical heart valve, previous VTE), iv) patient (or their delegate) is unable or unwilling to provide informed consent,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were admitted to hospital with COVID-19 or who contracted COVID-19 while in hospital and discharged to anywhere but an acute care hospital.
Sampling Method: Non-Probability Sample
Enrollment: 510 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
VTE | 90 days
  incidence of acute symptomatic VTE at 90 days after hospital discharge

SECONDARY OUTCOMES:
Risk for VTE | 90 days
  risk factors for VTE after hospital discharge (age, sex, D-dimer, duration of hospitalization, dose of prophylactic anticoagulation during hospitalization)

CONTACTS AND LOCATIONS:
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided